CLINICAL TRIAL: NCT05937464
Title: Effects of Robotic-Assisted Gait Training on Functional Independence, Functional Capacity, and Quality of Life in Patients With Stroke: A Randomized Controlled Study
Brief Title: Effects of Robotic-Assisted Gait Training in Patients With Stroke (EoRAGTiPwS)
Acronym: EoRAGTiPwS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/2021-66
Record Dates: First submitted 2023-05-16; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Stroke, Robotic Rehabilitation
Keywords: Stroke; Robotic Rehabilitation; Functional Independence; Functional Capacity; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exoskeleton ExoAthlet group (Experimental)
  Interventions: Other: Exoskeleton ExoAthlet group
- Lokomat Free-D group (Experimental)
  Interventions: Other: Lokomat Free-D group

INTERVENTIONS:
Other: Exoskeleton ExoAthlet group — This group included 16 patients who had stroke. The patients was evaluated with Functional Independence Measure (FIM), physical function with 30-second chair stand test (30-CST), functional capacity with 6-Minute Walk Test (6MWT), and their quality of life with Short Form 36 (SF36). Conventional physiotherapy program was applied to groups for eight weeks, three days a week, each session 60 minutes. Then, one group received walking exercise training with exoskeleton ExoAthlet (ExoAtlet 1 model/2019, Russia). Participants were assessed at baseline and post-intervention.
  Arms: Exoskeleton ExoAthlet group
Other: Lokomat Free-D group — This group included 16 patients who had stroke. The patients was evaluated with Functional Independence Measure (FIM), physical function with 30-second chair stand test (30-CST), functional capacity with 6-Minute Walk Test (6MWT), and their quality of life with Short Form 36 (SF36). Conventional physiotherapy program was applied to groups for eight weeks, three days a week, each session 60 minutes. Then, one group received walking exercise training with Lokomat Free-D (Hocoma, Lokomat Pro Free-D model/2015, Switzerland). Participants were assessed at baseline and post-intervention.
  Arms: Lokomat Free-D group

SUMMARY:
This study was conducted to examine effects of gait training with exoskeleton ExoAthlet and Lokomat Free-D on functional independence, functional capacity and quality of life in stroke patients.

DETAILED DESCRIPTION:
The study included 32 patients who had stroke. Participants were randomized into two groups. Functional independence of patients was evaluated with Functional Independence Measure (FIM), physical function with 30-second chair stand test (30-CST), functional capacity with 6-Minute Walk Test (6MWT), and their quality of life with Short Form 36 (SF36). Conventional physiotherapy program was applied to groups for eight weeks, three days a week, each session 60 minutes. Then, one group received walking exercise training with exoskeleton ExoAthlet (ExoAtlet 1 model/2019, Russia), other group with Lokomat Free-D (Hocoma, Lokomat Pro Free-D model/2015, Switzerland). Participants were assessed at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between18-65 years old
* Patients who had a stroke at least three months ago
* Can independently ambulated

Exclusion Criteria:

* Heart failure and rhythm disorder,
* Visual and cognitive problems,
* Neglect phenomenon (Neglect Syndrome),
* Cerebellar pathology,
* Any lower extremity surgery
* An additional neurological pathology that could prevent receiving a training program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | At baseline
  : Participants' functional independence was assessed with the Turkish version of the Functional Independence Measure (FIM).17 FIM indicates the degree of independence of an individual in basic physical and cognitive activities in daily life. FIM consists of 18 questions and basically measures 2 parameters: 1) physical/motor function, 2) cognitive/cognitive function. Each item is scored at 7 levels (1-7), with 'level 1' representing full dependance and 'level 7' completely independence. The FIM total score is between 18-126 points. The higher the score an individual gets, the higher the level of independence means. FIM is the most preferred and used activity scale in the field of rehabilitation.
30-Second chair stand test | At baseline
  The physical functionality of the participants was assessed with the 30-Second chair stand test.18 The 30-second chair stand test (30-CST) is a measure of lower body strength and endurance. Participants were asked to sit in a standard-height chair (with a seat height of 43 cm) with arms crossed over the chest, then stand fully and sit down again as many times as possible within 30 s. In order to decrease the effect of learning, all tests began with three to five practices.
6- Minute walk test | At baseline
  The functional capacities of the participants were evaluated with the 6-Minute Walk Test (6MWT), which can determine the functional capacity of individuals with a single measurement in neurological diseases.19 In the study, a 30 m long straight line was divided into 3 m intervals and the total distance walked at the end of 6 minutes was calculated. Rest period of 10 minutes was given before the test. The importance of the distance to be walked was emphasized to the individuals participating in the study and they were asked to walk as fast as they could without running. At the end of the test, the distance that the individuals could walk was recorded in meters (m).
36-Item Short Form Health Survey | At baseline
  The quality of life of the participants was evaluated with the Turkish version of the Medical Outcomes 36-Item Short Form Health Survey (SF-36) scale.20 SF-36 is a 36-item self-assessment scale consisting of eight sub-parameters. This scale consists of Physical functioning, Role limitations: Physical/Emotional, Social functioning, Mental health, Vitality, General health perception sub-parameters. Each subscale is scored between 0-100. An increase in the score indicates an improvement in the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Private rehabilitation center in Istanbul, Istanbul, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No